CLINICAL TRIAL: NCT02835248
Title: A Novel System to Detect Falls in Real-life Conditions
Status: Completed | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: Brigham and Women's Hospital (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 15-0930-01
Record Dates: First submitted 2016-07-08; First posted 2016-07-18 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Falls

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: Older adult study participants will be recruited from the cohort of participants in the STRIDE Study at the Boston trial site (http://www.stride-study.org/).
  Interventions: Other: Fall Detection

INTERVENTIONS:
Other: Fall Detection — All participants will wear a device configured to detect falls.
  Other Names: ActivePERS

SUMMARY:
Medical alert devices with automatic fall detection functionality use accelerometry to detect a fall and can signal for help if the wearer forgets to, or is incapable of, pressing the alert button. This can save lives and prevent complications associated with long periods of time spent on the floor after a fall. In this project, the sensitivity and false alarm rate of a commercially available medical alert device will be tested in a population of 200 community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the STRIDE Study at the Boston trial site (http://www.stride-study.org/).

Exclusion Criteria:

* Uses a medical alert device

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older adult study participants will be recruited from the cohort of participants in the STRIDE Study at the Boston trial site (http://www.stride-study.org/).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The sensitivity and specificity of ActivePERS fall detection algorithms will be measured by comparing the occurence of falls detected by the wearable device to study participant self reported falls | 2 years

SECONDARY OUTCOMES:
Near falls as measured by patient self report | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shalendar Bhasin, MD, Principal Investigator — Brigham and Women's Hospital; Joseph T Gwin, PhD, Principal Investigator — BioSensics; Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No